CLINICAL TRIAL: NCT02377232
Title: Simultaneous Improvement in Colon Cancer Screening Rates and Patient-Centered Care
Acronym: CRCSreening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Screening
Other Study IDs: 14-1976
Record Dates: First submitted 2015-02-25; First posted 2015-03-03 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Outreach for Colon Cancer Screening (Active Comparator): Receives standard of care outreach concerning colon cancer screening.
  Interventions: Behavioral: Usual Care Outreach for Colon Cancer Screening
- Decision Aid for Colon Cancer Screening (Active Comparator): Receives colon cancer screening decision aid intervention in addition to outreach.
  Interventions: Behavioral: Decision Aid for Colon Cancer Screening

INTERVENTIONS:
Behavioral: Decision Aid for Colon Cancer Screening — Paper decision aid describing different screening options for colon cancer
  Arms: Decision Aid for Colon Cancer Screening
Behavioral: Usual Care Outreach for Colon Cancer Screening — Patients overdue for colon cancer screening are contacted and outreach is performed in an effort to schedule colonoscopy
  Arms: Usual Care Outreach for Colon Cancer Screening

SUMMARY:
Several screening methods exist to screen patients for CRC ranging from invasive (i.e., colonoscopy) to less invasive (i.e., testing the stool for blood). Although choice between screening methods is recommended, patients are not currently offered an unbiased choice and physicians generally recommend only colonoscopy. In this project, the investigators will answer the following questions: 1) Is it feasible to incorporate a DA in the AHP protocol?; 2) Is it feasible to incorporate mailing patients a stool blood test?; 3) Does the DA change CRC screening decision quality, using proxy measures such as knowledge and intent; and 4) Does the DA change the proportion of participants that complete a CRC screening test? To answer these questions the investigators will compare survey responses and CRC test type completed between two AHP CRC surveillance patients groups - those that received usual care versus those that received the DA.

DETAILED DESCRIPTION:
At the University of Colorado Hospital primary care clinics, only 59% of eligible patients are up to date with current colorectal cancer (CRC) screening. This is below the national average of 65% and well below the healthy people 2020 goal of 70.5%. Several screening methods exist to screen patients for CRC ranging from invasive (i.e., colonoscopy) to less invasive (i.e., testing the stool for blood). Although choice between screening methods is recommended, patients are not currently offered an unbiased choice and physicians generally recommend only colonoscopy. Further, the investigators know from research that choice increases screening rates. Unfortunately, many people do not follow through when only colonoscopy is offered. However, participants in one study were nearly twice as likely to be screened if they were offered a choice between colonoscopy and fecal occult blood testing rather than being offered colonoscopy alone. Thus, in this project, the investigators aim to examine the feasibility of incorporating a patient decision aid (DA) for patients in CRC screening surveillance with the Ambulatory Health Promotion (AHP) using a pre/post design. The investigators will answer the following questions: 1) Is it feasible to incorporate a DA in the AHP protocol?; 2) Is it feasible to incorporate mailing patients a stool blood test?; 3) Does the DA change CRC screening decision quality, using proxy measures such as knowledge and intent; and 4) Does the DA change the proportion of participants that complete a CRC screening test? To answer these questions the investigators will compare survey responses and CRC test type completed between two AHP CRC surveillance patients groups - those that received usual care versus those that received the DA.

ELIGIBILITY:
Inclusion Criteria:

* Individuals that fall within the age range for CRC screening surveillance (age 50 to < = 75 years) from AHP
* Are eligible for CRC screening surveillance from AHP
* Were seen in the last 18 months by a provider at one of the primary medical care clinics from the University of Colorado General Internal Medicine, Family Medicine, or the Women's Integrated Services in Health clinic, and the individual's primary medical care provider has provided approval for AHP CRC outreach to an AHP staff person
* Have no record of a colonoscopy within the last 10 years,
* Have no record of flexible sigmoidoscopy or double-contrast barium enema within the past 5 years, or
* Have no record of FOBT within the past year.

Exclusion Criteria:

* Individuals that do not speak English
* Individuals that have limited cognitive function/developmental disabilities
* Individuals that have a personal or family history of CRC (previous adenomatous polyp), and/or, have a signs and symptoms colonoscopy order from their primary care physician
* Not eligible for CRC screening surveillance from AHP
* Have a terminal medical illness that would otherwise categorize them as inappropriate candidates for CRC screening as noted in their EPIC EMR:
* The individual exhibits any of the following:

  * personal history of CRC, colectomy, colostomy, or ileostomy; currently prescribed anti-coagulation medications (ReoPro (abciximab), Aggrenox (aspirin plus dipyridamole), Persantine (dipyridamole), Integrilin (eptifibatide), Ticlid (ticlopidine), Aggrastat (tirofiban), Heparin, Coumadin (warfarin), Pradaxa (dabigatran), Xarelto (rivaroxaban)); currently prescribed plavix (clopidogrel); on chronic oxygen; have end-stage renal disease; have unstable angina; have arrhythmia/atrial fibrillation; have cardiomyopathy; currently weighs >350 pounds; have cystic fibrosis; and/or, are insured by the Colorado indigent care program (CICP) or Medicaid-Old age pension, AARP Medicare/Secure Horizons (except PFFS), Denver Health Managed Medicaid, Evercare; Kaiser (not the prescriber of origin), Medicare Complete, New Medicaid, New CICP. Furthermore, dependent on the severity of the condition, the following are gauged for exclusion criteria and noted in the AHP CRC screening surveillance test notes to then inquire about appropriate candidacy for a colonoscopy: diabetes mellitus (insulin, oral, or both), chronic obstructive pulmonary disease, emphysema, reactive airway disease; chronic renal disease; multiple sclerosis; seizure disorder; murmurs; hepatitis; human immunodeficiency virus /acquired immunodeficiency syndrome ; congestive heart failure; coronary artery disease; aortic aneurysm; history of coronary artery bypass graft; heart valve issues (prolapse, regurgitation, etc.); tachycardia; bradycardia; history of myocardial infarction.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Colon Cancer Screening Intent | 6 months
  Measured using a survey instrument to assess intent

SECONDARY OUTCOMES:
Colon Cancer Screening Completed | 6 Months
  Measured through retrospective chart reviews to check for completed screening

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Lewis, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No